CLINICAL TRIAL: NCT02795299
Title: Phase 2, Rand, Placebo-Controlled, Double-Blind, Dose Ranging Study to Evaluating Safety/Efficacy of Gerilimzumab in Patients With Moderately to Severely Active Rheumatoid Arthritis Inadequately Treated With Methotrexate or TNFα Antagonist
Brief Title: Study Evaluating Gerilimzumab´s Safety/Efficacy for Patients MTX or TNFα Antagonist Failed in Rheumatoid Arthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not started due to Sponsor decision to not move forward with compound.
Sponsor: Bird Rock Bio, Inc. (Industry)
Collaborators: Techtrials Pesquisa e Tecnologia Ltda (Unknown); Pharmagenix (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRB-008-003
Record Dates: First submitted 2016-05-02; First posted 2016-06-10 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Gerilimzumab 5/2 mg/Methotrexate/folate (Active Comparator): • 5 mg gerilimzumab loading dose followed by 2 mg gerilimzumab every 8 weeks + 15-25 mg Methotrexate every week + 1 mg folic acid once daily
  Interventions: Drug: Gerilimzumab; Drug: Methotrexate; Drug: Folic Acid
- Gerilimzumab 10/5mg/Methotrexate/folate (Active Comparator): • 10 mg gerilimzumab loading dose followed by 5 mg gerilimzumab every 8 weeks + 15-25 mg Methotrexate every week + 1 mg folic acid once daily
  Interventions: Drug: Gerilimzumab; Drug: Methotrexate; Drug: Folic Acid
- Gerilimzumab 20/10mg/Methotrexate/folate (Active Comparator): • 20 mg gerilimzumab loading dose followed by 10 mg gerilimzumab every 8 weeks + 15-25 mg Methotrexate every week + 1 mg folic acid once daily
  Interventions: Drug: Gerilimzumab; Drug: Methotrexate; Drug: Folic Acid
- Placebo/Methotrexate/folate (Placebo Comparator): • Placebo every 8 weeks + 15-25 mg Methotrexate every week + 1 mg folic acid once daily
  Interventions: Drug: Methotrexate; Drug: Folic Acid; Drug: Placebo

INTERVENTIONS:
Drug: Gerilimzumab — Either Gerilimzumab 5 mg followed by 2 mg, or Gerilimzumab 10 mg followed by 5 mg or Gerilimzumab 20 mg followed by 10 mg are to be administered once every 8 weeks during the treatment period of the study.
  Arms: Gerilimzumab 10/5mg/Methotrexate/folate; Gerilimzumab 20/10mg/Methotrexate/folate; Gerilimzumab 5/2 mg/Methotrexate/folate
Drug: Methotrexate — Methotrexate (MTX) to be administered once a week every week during the treatment period.
Drug: Folic Acid — Acid folic (folate) 1mg to be administered once daily during the treatment period.
Drug: Placebo — 10 mM acetate, 9% (w/v) sucrose, and 0.006% (w/v) polysorbate 20 at pH 5.2 ± 0.3
  Arms: Placebo/Methotrexate/folate

SUMMARY:
Phase 2 Study Evaluating Gerilimzumab's Safety/Efficacy for Patients with an Inadequate Response to MTX or a TNFα Antagonist in Rheumatoid Arthritis.

DETAILED DESCRIPTION:
The trial will include adult patients 18-80 years of age with active disease who have demonstrated an inadequate response to treatment with MTX. Eligible patients will enter a 6-week screening period receiving 15-25 mg MTX QWK (patients will remain on their current dose and route of administration of MTX through the screening period). Patients on a dose of MTX less than 15mg QWK will have their dose of MTX increased to 15mg QWK at the initial screening visit) followed by randomization in a 1:1:1:1 ratio to 1 of 3 doses of gerilimzumab (5, 10, or 20 mg loading dose followed by 2 mg, 5 mg or 10 mg of gerilimzumab Q8W) plus MTX, or placebo plus MTX for 12 weeks of treatment. Gerilimzumab and placebo will be administered as SC injections Q8W; MTX will continue to be administered as by same route of administration (tablets, SC, or IM injection) QWK.

ELIGIBILITY:
Key Inclusion Criteria

Each patient must meet the following inclusion criteria to be enrolled in the study:

1. Men or women, ages 18 to 80 years, inclusive;
2. Diagnosis of moderately to severely active RA for at least 3 months prior to screening as according to 2010 EULAR/ACR classification criteria for at least 3 months prior to screening with ACR functional class I-III;
3. Have active RA with ≥4 swollen and ≥4 tender joints (28 joint count) throughout the screening period (all visits) and baseline visit at Week 0 baseline. Must meet above criteria in order to enter screening phase at all screening visits to be randomized;
4. Current treatment with stable dose of oral MTX (i.e., 15-25 mg/week for >6 weeks) prior to screening. Patients will remain on their current dose and route of administration of MTX through the screening period. Patients must also remain on a stable dose and route of administration of MTX and folic acid supplementation throughout the randomized treatment phase of the study. Patients on a dose of MTX <15 mg QWK may have their dose of MTX increased to 15mg QWK at the initial screening visit providing that they meet all other entry criteria;
5. Demonstrated an inadequate response to previous or current MTX treatment and/or a single TNFα inhibitor;
6. C-reactive Protein (CRP) above the ULN for the central laboratory at the time of screening;
7. Positive Cyclic Citrullinated Peptide (CCP) antibody or Rheumatoid Factor (RF) from the central laboratory at the screening visit;
8. Previous treatment with a single TNFα antagonist is permitted, providing there has been:

   * An inadequate response to an approved or investigational: TNFα antagonist despite completing an induction regimen with any approved or experimental TNFα antagonist per the current labeling, study protocol or institutional standard of care
   * Recurrence of symptoms during maintenance dosing with a TNFα antagonist following prior clinical benefit(discontinuation despite clinical benefit does not qualify)
   * History of intolerance to a TNFα antagonist (including but not limited to infusion or injection related reaction, demyelination, congestive heart failure or serious infection)
9. Considered to be in stable health in the opinion of the Investigator, as determined by:

   * A pre-study physical examination with no clinically significant abnormalities aside from those related to rheumatoid disease
   * Vital signs (VS): heart rates at screening must be ≥ 50 bpm; and systolic blood pressure (SBP) and diastolic blood pressure (DBP) ≥ 90 and ≥ 55, respectively at all screening visits
   * Liver function tests (ALT/AST, bilirubin and Alkaline phosphatase) <2X the upper limit of normal) at all screening visits
10. Subject is not pregnant (negative pregnancy test) or nursing and is not planning pregnancy or initiation of breast-feeding over the duration of the study
11. Women of child-bearing potential must use effective contraception for the duration of the study until 180 days after study treatment discontinuation
12. Men who have sexual relationships with women of child-bearing potential will agree to use an effective means of contraception for the duration of the study until 60 days after study treatment discontinuation. In addition, men must agree not to donate sperm for the duration of the study until 60 days after study treatment discontinuation.

Key Exclusion Criteria

1. History of an autoimmune disease other than RA or with significant systemic involvement secondary to RA. Patients with a history of diabetes and or thyroiditis are eligible to participate if all other inclusion/exclusion criteria are met.
2. Diagnosis of any other arthritis (e.g., psoriatic arthritis or ankylosing spondylitis)
3. Secondary, non-inflammatory type of arthritis (e.g., osteoarthritis or fibromyalgia) that in the Investigator's opinion could interfere with the evaluation of the effect of study medication on the subjects primary diagnosis of RA

   Concomitant medication/therapy exclusions:
4. Have received approved or investigational biological or targeted synthetic DMARD therapies for RA (except TNFα inhibitors (as described above) prior to screening;
5. Any prior exposure to natalizumab, efalizumab, rituximab, tocilizumab, or abatacept, or tofacitinib or any other Janus kinase [JAK]-inhibitors, or anti IL-1 therapies;
6. Within 30 days prior to enrollment, have received any of the following for the treatment of underlying disease:

   - Non-biologic therapies (e.g., cyclosporine, tacrolimus, thalidomide)
7. Have received prior approved or Investigational therapy blocking the interleukin-6 (IL-6) pathway, at any time
8. Have received any live (includes attenuated) vaccination within 60 days prior to screening (e.g., injectable influenza and pneumococcal vaccines are allowed, but nasal influenza vaccine is not) or anticipate needing any such vaccines for the duration of the study until 30 days after study treatment discontinuation
9. Subject has previously received any other investigational (either approved or unapproved) drug within 30 days or 5 half-lives (whichever is longer) prior to the screening visit
10. History of tuberculosis (patients with previous TB treated with local standard of care and with documentation of completion of this therapy will be allowed)
11. Any identified congenital or acquired immunodeficiency (e.g., common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation)
12. Positive for Hepatitis BSAg or Hepatitis C virus
13. Infection requiring hospitalization or intravenous antimicrobial therapy, or opportunistic infection within 4 weeks of screening with last dose of antibiotics received within 2 weeks of screening
14. History of malignancy within the 5 years prior to Screening except for adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
15. History of diverticulitis, diverticulosis, or intestinal perforation
16. History of anaphylactic reactions to biologic therapy requiring medical attention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean DAS28-CRP (Disease Activity Score 28 using the C-Reactive Protein value) | to be applied in weeks - 6, -2, -1, 0, 4, 8, 12 and 16

SECONDARY OUTCOMES:
The proportion of patients meeting the ACR20 (American College of Rheumatology 20%) response criteria at Week 12 | to be applied in weeks -6, 0, 4, 8, 12 and 16

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Keiserman, Principal Investigator — LMK - Serviços Medicos Sociedade Simples, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Result] Pereira IA, Mota LM, Cruz BA, Brenol CV, Fronza LS, Bertolo MB, Freitas MV, Silva NA, Louzada-Junior P, Giorgi RD, Lima RA, Pinheiro Gda R; Brazilian Society of Rheumatology. 2012 Brazilian Society of Rheumatology Consensus on the management of comorbidities in patients with rheumatoid arthritis. Rev Bras Reumatol. 2012 Aug;52(4):474-95. English, Portuguese. PMID 22885417
- [Result] McInnes IB, Schett G. The pathogenesis of rheumatoid arthritis. N Engl J Med. 2011 Dec 8;365(23):2205-19. doi: 10.1056/NEJMra1004965. No abstract available. PMID 22150039
- [Result] Smolen JS, Weinblatt ME, Sheng S, Zhuang Y, Hsu B. Sirukumab, a human anti-interleukin-6 monoclonal antibody: a randomised, 2-part (proof-of-concept and dose-finding), phase II study in patients with active rheumatoid arthritis despite methotrexate therapy. Ann Rheum Dis. 2014 Sep;73(9):1616-25. doi: 10.1136/annrheumdis-2013-205137. Epub 2014 Apr 3. PMID 24699939
- [Result] Mease P, Strand V, Shalamberidze L, Dimic A, Raskina T, Xu LA, Liu Y, Smith J. A phase II, double-blind, randomised, placebo-controlled study of BMS945429 (ALD518) in patients with rheumatoid arthritis with an inadequate response to methotrexate. Ann Rheum Dis. 2012 Jul;71(7):1183-9. doi: 10.1136/annrheumdis-2011-200704. Epub 2012 Feb 10. PMID 22328739